CLINICAL TRIAL: NCT03991949
Title: Evaluation of Preterm Infants Fed Post-Discharge Preterm Infant Formula With Prebiotic
Brief Title: Evaluation of Preterm Infants Fed Post-Discharge Preterm Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL35
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Infant Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Infant Formula (Experimental): Ready-to-feed, milk-based formula
  Interventions: Other: Experimental Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Formula fed Ad libitum

SUMMARY:
This single-group study will assess growth and tolerance of infants fed a post-discharge preterm infant formula containing a prebiotic.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth less than 37 weeks
* Birth weight less than 3200 g (approximately 7 pounds)
* Postmenstrual age is 34 0/7 through 41 0/7 weeks at enrollment
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study
* The currently-fed formula is a milk-based infant formula at a caloric density of ≤ 24 Cal/fl oz.
* Singleton, twin, or triplet births only.
* Parent(s) confirm their intention not to administer solid foods or juices to their infant from enrollment through the duration of the study, unless instructed otherwise by their healthcare professional.
* Participant's parent(s) has voluntarily signed and dated an ICF, approved by an IRB/IEC and provided HIPAA (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Participant is taking and plans to continue taking medications, home remedies, herbal preparations, prebiotics or probiotics, rehydration solutions, or parenteral nutrition
* Participant is known to require elective surgery with hospitalization, other than uncomplicated outpatient surgery, during the course of the study.
* Participant is in another study that has not been approved as a concomitant study
* Participant has an allergy or intolerance to any ingredient in the study product
* Participant is currently receiving oxygen therapy
* Participant is currently receiving antibiotics
* Participant is currently receiving tube feedings

Ages: 34 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Weight | SDAY 1 to SDAY 56
  Change in weight-for-age z-score

SECONDARY OUTCOMES:
Stool Characteristics | Study Day (SDAY) 1 to SDAY 56
  Parent completed diary
Formula Intake | SDAY 1 to SDAY 56
  Parent completed diary
Length | SDAY 1 to SDAY 56
  Interval length gain per day
Head Circumference | SDAY 1 to SDAY 56
  Interval HC gain per day

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Johnson, RDN, LD, Study Chair — Abbott Nutrition
Locations (7):
- United States (7):
  - University of South Florida, Tampa, Florida
  - University of Louisville Research Foundation, Inc., Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Women's Hospital at Renaissance - Doctors Hospital at Renaissance, Edinburg, Texas
  - Maximos Ob/Gyn, League City, Texas

IPD SHARING:
Plan to Share IPD: No